CLINICAL TRIAL: NCT00380731
Title: fMRI of Emotional Reactivity Cognitive Regulation and CBT for Social Phobia
Brief Title: Effect of Behavior Therapy on Responses to Social Stimuli in People With Social Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James J. Gross, professor of psychology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH076074 (NIH); R01MH076074 (NIH); DATR A3-NSS
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Social Phobia
Keywords: Social Anxiety Disorder; Magnetic Resonance Imaging; Cognitive Behavior Therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive immediate cognitive behavioral therapy
  Interventions: Behavioral: Individual Cognitive Behavioral Therapy
- 2 (Experimental): Participants will receive cognitive behavioral therapy with a 16-week delayed start
  Interventions: Behavioral: Individual Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Individual Cognitive Behavioral Therapy — CBT includes 16 weekly 60-minute individual CBT sessions for social anxiety disorder.

SUMMARY:
This study will evaluate the effect of cognitive behavioral therapy on the brain during emotional and behavioral responses to social stimuli in people with social phobia.

DETAILED DESCRIPTION:
Social phobia, also known as social anxiety disorder, is a common, often debilitating condition. People with social phobia experience high levels of anxiety when they participate in social situations or perform in front of others. Approximately 80% of social phobia cases occur before the age of 18, and often precede other anxiety, mood, and substance abuse or dependence disorders. Physical symptoms typically accompany the intense anxiety caused by the disorder, and may include blushing, profuse sweating, trembling, nausea, and difficulty talking. Cognitive-behavioral therapy (CBT) has been shown to be an effective treatment method for most people with social phobia. Approximately 30% of people with the disorder, however, do not respond to CBT treatment. A better understanding of the neural mechanisms underlying social phobia and CBT's effect on these mechanisms will help physicians to better predict the best treatment for different patients. This study will evaluate the effect of CBT on how the brain processes emotional and behavioral responses to social stimuli in people with social phobia.

Participants in this open-label study will be randomly assigned to either immediate or delayed treatment with CBT. Participants who are assigned to immediate CBT will attend 16 sessions of individual CBT immediately following baseline assessments. Participants assigned to the delayed treatment condition will begin attending CBT sessions approximately 5 months following baseline assessments. Outcomes will be assessed for all participants at baseline, immediately post-treatment, and at Months 5 and 10 post-treatment. An fMRI scan will be used to measure neural responses to social stimuli, and various questionnaires and scales will be used to assess anxiety symptom severity. Participants in the delayed treatment group will be assessed on one additional occasion before they begin treatment after the 5-month waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for generalized social phobia
* English-speaking
* Eligible to participate in fMRI scanning
* Willing to use an effective form of contraception throughout the study

Exclusion Criteria:

* Currently undergoing any psychotherapy or pharmacotherapy (e.g, selective serotonin reuptake inhibitors, benzodiazepines, beta-blockers, anti-psychotics, blood thinners, thyroid hormone influencing agents, diabetic medications, or anticonvulsants)
* History of neurological or cardiovascular disorders, brain surgery, electroconvulsive or radiation treatment, brain hemorrhage or tumor, stroke, seizures or epilepsy, diabetes, hypo- or hyperthyroidism, or head trauma with loss of consciousness for more than 5 minutes
* Smokes cigarettes daily
* History of or current diagnosis of schizophrenia, schizoaffective disorder, organic mental disorder, bipolar disorder, or antisocial, schizotypal, or schizoid personality disorders
* Suicidal thoughts
* Clinically significant and/or unstable medical disease
* Pregnant or breastfeeding
* Alcohol or substance abuse or dependence within the 12 months prior to study entry
* History of or current seizure disorder (except febrile seizure disorder during childhood)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | Measured at Months 4, 7, 10, 13, and 16
fMRI BOLD response | Measured at Month 4
Behavioral assessment | Measured at Months 4 and 16

SECONDARY OUTCOMES:
Clinical Global Impression Improvement Scale | Measured at Months 4 and 16
Social Interaction Anxiety Scale | Measured at Months 4, 10, and 16
Sheehan Disability Scale | Measured at Months 4, 10, and 16
Quality of Life Inventory | Measured at Months 4, 10, and 16

CONTACTS AND LOCATIONS:
Overall Officials: James J. Gross, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Butler RM, O'Day EB, Kaplan SC, Swee MB, Horenstein A, Morrison AS, Goldin PR, Gross JJ, Heimberg RG. Do sudden gains predict treatment outcome in social anxiety disorder? Findings from two randomized controlled trials. Behav Res Ther. 2019 Oct;121:103453. doi: 10.1016/j.brat.2019.103453. Epub 2019 Aug 9. PMID 31430688
- [Derived] Goldin PR, Ziv M, Jazaieri H, Weeks J, Heimberg RG, Gross JJ. Impact of cognitive-behavioral therapy for social anxiety disorder on the neural bases of emotional reactivity to and regulation of social evaluation. Behav Res Ther. 2014 Nov;62:97-106. doi: 10.1016/j.brat.2014.08.005. Epub 2014 Aug 21. PMID 25193002
- [Derived] Goldin PR, Lee I, Ziv M, Jazaieri H, Heimberg RG, Gross JJ. Trajectories of change in emotion regulation and social anxiety during cognitive-behavioral therapy for social anxiety disorder. Behav Res Ther. 2014 May;56:7-15. doi: 10.1016/j.brat.2014.02.005. Epub 2014 Feb 28. PMID 24632110
- [Derived] Ziv M, Goldin PR, Jazaieri H, Hahn KS, Gross JJ. Emotion regulation in social anxiety disorder: behavioral and neural responses to three socio-emotional tasks. Biol Mood Anxiety Disord. 2013 Nov 4;3(1):20. doi: 10.1186/2045-5380-3-20. PMID 24517388
- [Derived] Goldin PR, Ziv M, Jazaieri H, Hahn K, Heimberg R, Gross JJ. Impact of cognitive behavioral therapy for social anxiety disorder on the neural dynamics of cognitive reappraisal of negative self-beliefs: randomized clinical trial. JAMA Psychiatry. 2013 Oct;70(10):1048-56. doi: 10.1001/jamapsychiatry.2013.234. PMID 23945981